CLINICAL TRIAL: NCT00423969
Title: Galantamine Augmentation of Escitalopram for Treatment of Depression Associated Cognitive Impairment in Outpatients - A Randomized Single Blind Clinical Trial
Brief Title: Galantamine Augmentation of Escitalopram for Treatment of Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0301-35; 45-869-96
Record Dates: First submitted 2005-09-14; First posted 2007-01-18 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2007-01

CONDITIONS: Depression
Keywords: Depression; Cognitive Impairment
MeSH Terms: conditions — Depression; Cognitive Dysfunction | interventions — Galantamine; Escitalopram

INTERVENTIONS:
Drug: Galantamine
Drug: Escitalopram

SUMMARY:
The purpose of this study is to investigate whether the addition of galantamine to a commonly used antidepressant, escitalopram (Lexapro), will be useful in the treatment of memory and other thinking problems that are frequently seen in depression. At present, galantamine is approved for use in the treatment of Alzheimer's disease or dementia, but not for use for the treatment of depression in younger patients.

Possible genetic effects of depressed individuals will also be studied. This study is involved in collecting blood from patients with depression. DNA, the genetic material in our cells, will be obtained from these blood samples. The DNA will be studied to determine the contribution of different genes to the development of depression. These blood samples are extremely useful to researchers who are trying to determine the genetic risk factors that may lead to depression.

DETAILED DESCRIPTION:
HYPOTHESES/OBJECTIVES

Aim 1: To investigate whether patients treated with escitalopram in combination with galantamine will show a significantly greater improvement of depression compared to patients treated with escitalopram alone.

H1: Patients treated with escitalopram and galantamine combination will have significantly greater improvement on the Hamilton Depression Rating Scale (HDRS) and Clinical Global Improvement (CGI) scale compared to patients treated with escitalopram and placebo.

Aim 2: To investigate whether treatment with escitalopram in combination with galantamine will lead to a greater improvement of cognitive function in depressed patients compared to escitalopram alone.

H2: Patients treated with escitalopram and galantamine combination will have significantly greater improvement of scores on Selective Reminding Test (SRT) and Trail Making Test (TMT) than patients treated with escitalopram and placebo.

Study Design and Method:

This will be a randomized, single blind, parallel-group, placebo controlled study in which a total of 20 subjects, 10 in each arm: one arm would be escitalopram + galantamine treatment and the other arm will be escitalopram + placebo treatment. The subject will be blinded against the galantamine or placebo, but will be unblinded against escitalopram. The total duration of this study will be 10 weeks. After the baseline visit, patients will complete 8 weeks of the study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60 years of age inclusive
2. Satisfy DSM-IV-TR criteria for Major Depression
3. RAVLT scores decreased from normative mean for age
4. 17 item HDRS rating > 18
5. Give informed consent as approved by local IRB
6. On no antidepressants or wanting to be tapered off current antidepressant medication due to side effects or inefficacy; and
7. Not on monoamine oxidase inhibitors (MAOIs) for 3 weeks before start of the study.

Exclusion Criteria:

1. Comorbid psychotic disorder such as schizophrenia or schizoaffective disorder
2. Significant suicidal or homicidal risk
3. Clinically significant medical illness
4. Allergy or intolerance to escitalopram or galantamine
5. Woman of child bearing age (except if surgically sterile or have had tubal ligation)
6. Satisfy criteria for substance dependence within 6 months prior to start of the study
7. History of intolerance to escitalopram or galantamine; and
8. On any medication with significant adverse interaction with either escitalopram or galantamine.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2003-11; Study Completion 2005-09

PRIMARY OUTCOMES:
Decrease in depression symptoms measured by Hamilton Depression Rating Scale and Clinical Global Improvement Scale
Improvement of cognitive measures scores:Selective Reminding Test, Trail Making Test and others

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — university
Locations (1):
- IU Adult Psychiatric Clinic, Indianapolis, Indiana, United States